CLINICAL TRIAL: NCT06812806
Title: Correlation Between the Change in the Antero-posterior Diameter of the Pelvic Side and the Incidence of Post-partum Urinary Incontinence
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: APD.IUP
Record Dates: First submitted 2024-12-30; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Urinary Incontinence
Keywords: incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
During pregnancy, the strength of the pelvic floor muscles may decrease, which can lead to musculoskeletal changes that may facilitate the onset of urinary incontinence. The investigators decided to conduct this study firstly to analyze, through simple ultrasound indices, how the contractile capacity of the pelvic floor muscles affects postpartum urinary incontinence; secondly to study the correlation between the use of perineal gymnastics, the incidence of postpartum urinary incontinence, and the strength of floor contraction.

DETAILED DESCRIPTION:
As part of the gynecologic ultrasound that is routinely performed, a transperineal scan will be performed, at rest and during maximal contraction to measure the lower portion of the pelvic floor groove. I order tho achieve this, doctors will illustrate to participants first verbally and then with the visual aid of the ultrasound monitor, how to contract the pelvic floor muscles. Transperineal ultrasound is performed by placing the ultrasound probe covered by a sterile glove at the level of the labia majora. Such ultrasound does not involve internal investigations and is in no way painful. The duration of the additional ultrasound scan involves a few minutes. In addition, in order to assess the presence of typical symptoms of urinary incontinence, the participant will undergo a standardized validated questionnaire in the Italian language, called ICIQ-UI SF, consisting of a series of questions that will investigate the type of urinary incontinence, its severity and its impact on her quality of life in the four weeks prior to administration. After delivery, the participant's medical records will be consulted and some data regarding the participant (age, ethnicity, height, weight, BMI, parity, gestational age at the time of delivery), the delivery (duration of stage II labor, mode of delivery, any vagino-perineal laceration and its degree) and the newborn (weight and head circumference measurement) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or older
* completion of delivery by vaginal delivery, vaginal delivery with obstetric suction cup or cesarean section
* acquisition of informed consent form

Exclusion Criteria:

* presence of severe maternal complications (e.g., ongoing postpartum hemorrhage, severe sepsis, pulmonary embolism, heart failure).
* presence of clinically demonstrable vulvar or vaginal infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants who have given birth by vaginal delivery, obstetric suction, or cesarean section and who result exclusively in inpatient care during puerperium.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the correlation between the proportional change in antero-posterior diameter of the pelvic hiatus and the incidence of postpartum urinary incontinence | On the second day, after delivery
  Evaluation of the correlation between the proportional change (in percentage) in pelvic antero-posterior diameter (APD) between rest and maximal contraction of pelvic floor muscles and the incidence of postpartum urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Aly Mohamed Alaaeldin Kamaleldin Aly Youssef, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy